CLINICAL TRIAL: NCT00429663
Title: Study of Locked Plates Versus Intramedullary Nails in Distal Femur Fractures: A Multicenter Randomized Trial Comparing IM Nails and Plate Fixation (S.O.L.V.E.D)
Brief Title: A Multicenter Randomized Trial Comparing IM Nails and Plate Fixation in Distal Femur Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Paul Tornetta, III, M.D., Paul Tornetta,III,M.D, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25934
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Femoral Fractures
Keywords: distal femur; femur fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IM Nails (Other): Reamed, Interlocking Intramedullary Nail - Randomized treatment
  Interventions: Device: reamed, interlocking intramedullary nail
- Plate Fixation (Other): Locking Periarticular Plate - Randomized Treatment
  Interventions: Device: locking periarticular plate

INTERVENTIONS:
Device: reamed, interlocking intramedullary nail — Standard of care device for femur fracture repair
  Arms: IM Nails
Device: locking periarticular plate — Standard of care device for femur fractures
  Arms: Plate Fixation

SUMMARY:
This study looks at two (2) types of surgical treatments and hopes to answer the question, "which is the best way to surgically treat a distal femur fracture?" Both procedures being studied are standard of care (used routinely) and use FDA approved devices. All medical and surgical treatment will be the same for participants as non-participants.

DETAILED DESCRIPTION:
The study is a randomized controlled multicenter trial in which individuals sustaining a fracture of the supracondylar (metaphyseal) region of the distal femur will be operatively managed by one of two strategies. The first strategy involves fixation of the fracture with a reamed, interlocking intramedullary nail (Nail Group). The second treatment strategy involves open reduction and internal fixation of the fracture with a locking periarticular plate (Plate Group). The null hypothesis of the study is that there will be no difference in the two groups with respect to the primary and secondary outcome measures. To the degree possible, patients in the two groups will receive post-operative care according to the same standards and protocols.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Fracture of the metaphyseal distal femur with or without intra-articular extension and with or without a TKA
* Fracture requiring operative treatment amenable to either IM nail or plate
* Informed consent obtained
* Patient is English speaking

Exclusion Criteria:

* Fracture of the metaphyseal distal femur with intra-articular communition,
* Fracture with vascular injury (Gustillo Type IIIC injury) requiring repair,
* Pathological fracture,
* Known metabolic bone disease,
* Contralateral distal femur fractures (bilateral injury) or ipsilateral lower extremity injury that would compromise function of the knee
* Retained hardware or existing deformity in the affected limb that would complicate IM nailing or plating
* Symptomatic knee arthritis
* Soft tissue injuries compromising either treatment method with nail or plate
* Surgical delay greater than 3 weeks for closed fractures or 24 hours for open fractures
* Immunocompromised
* Unable to comply with postoperative rehabilitation protocols or instructions (i.e. head injured or mentally impaired)
* Current or impending incarceration
* Unlikely to follow-up in surgeon's estimation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-02; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta, M.D., Principal Investigator — Boston University
Locations (22):
- United States (22):
  - University of California - Davis, Sacramento, California
  - Tampa General Hospital, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worchester, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Mary's Hospital - Mayo Clinic, Rochester, Minnesota
  - Barnes Hospital, St Louis, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - New York Hospital for Joint Diseases, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma/ Health Science, Oklahoma City, Oklahoma
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Campbell Foundation, Memphis, Tennessee
  - Orthopaedic Specialty Associates Fort Worth, Fort Worth, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although 160 participants were enrolled into the study, only 156 were included in the participant flow because 2 were found ineligible after consent and 2 withdrew before fixation.
Period: Overall Study
Arm/Group | IM Nails | Plate Fixation
Started | 76 | 80
Completed | 40 | 41
Not Completed | 36 | 39
Not completed — Lost to Follow-up | 24 | 31
Not completed — Physician Decision | 6 | 3
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Death | 4 | 0

BASELINE CHARACTERISTICS:
Population: 156 Patients were randomized to locked plate (80) or IM nail (76). Data for only 126 participants were captured due to patient withdrawal or incomplete data from sites
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Nails | Plate Fixation | Total
Number analyzed (Participants) | 58 | 68 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 41 | 48 | 89
  >=65 years | 16 | 20 | 36
Age, Continuous [Mean (Full Range); unit: years] | 51 [16 to 90] | 53 [19 to 90] | 51 [16 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 33 | 55
  Male | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: EQ-5D
Description: EQ-5D (EuroQol) Health Index taken at 3 months, 6 months, 12 months follow up. The EQ-5D measures the subjects health status in 5 categories (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and totals them into 1 score. Scoring ranges from 0-100, 100 being best.
Time Frame: 3 months, 6 months, 12 months
Population: 160 subjects were enrolled, but due to patient withdrawal or incomplete data from sites, only 126 subjects were followed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Nails | Plate Fixation
Number analyzed (Participants) | 58 | 68
units on a scale
  3 months | 69.23 (17.64) | 72.81 (18.85)
  6 months | 74.24 (13.65) | 73.04 (24.11)
  12 months | 79.07 (16.01) | 71.9 (23.34)

2. Primary Outcome: Short Musculoskeletal Functional Assessment (SMFA) Score
Description: The Short Musculoskeletal Functional Assessment (SMFA) score. The questionnaire consists of four categories: Daily Activities, Emotional Status, Arm and Hand Function, Mobility. All categories are scored together, totaling between 0-100. The lower the score, the better the subjects function.
Time Frame: 3 months, 6 months, 12 months
Population: 160 subjects were enrolled, but due to patient withdrawal or incomplete data from sites, only 126 subjects entered were followed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Nails | Plate Fixation
Number analyzed (Participants) | 58 | 68
units on a scale
  3 months | 38.76 (19.21) | 41.58 (19.17)
  6 months | 29.82 (18.79) | 31.92 (22.22)
  12 months | 22.18 (15.54) | 26.83 (23.18)

3. Primary Outcome: EQ Index
Description: EQ Index is a visual analog scale that the subject uses to rank overall health and wellness on a scale of 0.00-1.00, 1.00 being best.
Time Frame: 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Nails | Plate Fixation
Number analyzed (Participants) | 58 | 68
units on a scale
  3 months | 0.63 (.23) | 0.59 (.19)
  6 months | 0.73 (.27) | 0.68 (.20)
  12 months | 0.76 (.23) | 0.70 (.17)

4. Primary Outcome: SMFA - Bother Index
Description: The Bother Index is part of the SMFA. This section focuses on how much the injury is bothering the subject in terms of daily activities and use of injured area. The index totals are between 0-100. The lower the score, the less bothered the subject is by their injury.
Time Frame: 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Nails | Plate Fixation
Number analyzed (Participants) | 58 | 68
units on a scale
  3 months | 40.46 (21.95) | 36.75 (18.85)
  6 months | 28.23 (18.34) | 29.94 (24.34)
  12 months | 22.97 (19.12) | 28.93 (28.68)

5. Secondary Outcome: Valgus of Over 5 Degrees
Description: Valgus is a deformity involving oblique displacement of part of a limb away from the midline.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IM Nails | Plate Fixation
Number analyzed (Participants) | 58 | 68
participants | 10 | 20

ADVERSE EVENTS:
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months, 12 months
Arm/Group | IM Nails | Plate Fixation
Serious Adverse Events (participants affected / at risk) | 3/76 | 4/80
Other Adverse Events (participants affected / at risk) | 16/76 | 14/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM Nails (N=76) | Plate Fixation (N=80)
Subject expired due to cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subject expired due to cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Subject expired due to unknown reason (Cardiac disorders) | 1 (1) | 0 (0) — no information provided
Nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM Nails (N=76) | Plate Fixation (N=80)
Painful Implant (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7)
Pulmonary Embolism (Cardiac disorders) | 2 (2) | 1 (1)
Construct loosening (Surgical and medical procedures) | 4 (4) | 0 (0)
Deep Vein Thrombosis (Surgical and medical procedures) | 0 (0) | 2 (2)
Infection (Surgical and medical procedures) | 3 (3) | 2 (2)
Fractured Implant (Surgical and medical procedures) | 0 (0) | 1 (1)
Hardware Irritation (Surgical and medical procedures) | 0 (0) | 1 (1)
Contralateral TKA (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No